CLINICAL TRIAL: NCT04632342
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled, Phase 2a Clinical Trial to Evaluate the Efficacy and Safety of HL301 Versus Placebo on Radiation Pneumonitis in Unresectable Non-small Cell Lung Cancer Patients Treated With Curative Concurrent Chemoradiotherapy Using Paclitaxel and Carboplatin
Brief Title: Phase 2a Clinical Trial to Evaluate the Efficacy and Safety of HL301 on Radiation Pneumonitis in Non-small Cell Lung Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HL_HL301_203
Record Dates: First submitted 2020-11-13; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Radiation Pneumonitis; Lung Cancer
MeSH Terms: conditions — Radiation Pneumonitis; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): HL301 1,200mg/day
  Interventions: Drug: HL301 tablet 300mg
- Experimental group 2 (Experimental): HL301 1,800mg/day
  Interventions: Drug: HL301 tablet 300mg
- Control group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo of HL301 tablet

INTERVENTIONS:
Drug: HL301 tablet 300mg — * Experimental group 1 : 2 tablets at once, twice a day
  * Experimental group 2 : 2 tablets at once, three times a day
  Arms: Experimental group 1; Experimental group 2
Drug: Placebo of HL301 tablet — 2 tablets at once, three times a day
  Arms: Control group

SUMMARY:
The purpose of this clinical trial is to evaluate the safety when HL301 is administered to unresectable non-small cell lung cancer patients who receive chemoradiotherapy with Paclitaxel and Carboplatin and to search for a clinically appropriate dose by evaluating the efficacy by comparing the radiation pneumonia incidence rate with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, age ≥ 19 years
* Stage III non-small cell lung cancer(NSCLC) patient who without surgical treatment
* Patients scheduled for curative concurrent chemoradiotherapy

  * chemotherapy : paclitaxel and carboplatin
  * radiation therapy : IMRT, total 60~70Gy
* Eastern Cooperative Oncology Group(ECOG) performance status of 0 to 2 at the screening visit
* Subject whose remaining life expectancy is more than 6 months according to the judgment of investigator
* Volunteer, be willing and able to provide written informed consent for the trial

Exclusion Criteria:

* Subjects with pleural effusion
* Subjects with a weight loss of 10% or more within the last 6 months from the screening visit
* Subjects with a history of thoracic or neck radiotherapy or chemotherapy prior to screening visit
* Subjects with distant metastases
* Subjects with liver/renal dysfunction according to the following criteria on the screening test

  * Total Bilirubin >1.5 mg/dL
  * ALT or AST level is 2.0 times higher than the upper limit of normal (based on the institution)
  * Serum Creatinine >1.5 mg/dL
* Subjects with serious cardiovascular disease within 3 months prior to the screening visit (ex. arrhythmia, congestive heart failure, infarction, unstable angina etc)
* Subjects with serious systemic infection (≥ Grade 3, evaluated by CTCAE v5.0)
* Patients with chronic or interstitial lung disease (excluding patients with chronic obstructive pulmonary disease (COPD)), patients with chronic bronchitis, patients with pneumonia
* Subjects with thyroid dysfunction as present illness at the screening visit
* Subjects who administered systemic steroids within 4 weeks prior to the date of randomization (except for cases when administered to prevent hypersensitivity reaction of paclitaxel)
* Subjects who are hypersensitive to investigational products and standard anticancer treatments
* Subjects who participate in other clinical trials within 30 days prior to the screening visit and administer investigational drugs or apply clinical trial medical devices
* Women of childbearing age or men who do not agree to use a medically accepted method of contraception during the clinical trial
* Pregnant or breast-feeding
* Subjects who have clinical significance that is considered inappropriate for this clinical trial as judged by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with radiation pneumonia of ≥ Grade 2 | up to 24 weeks after completion of radiotherapy
  Percentage of subjects with radiation pneumonia of ≥ Grade 2 evaluated by CTCAE v5.0

SECONDARY OUTCOMES:
The incidence of radiation pneumonia | p to 24 weeks after completion of radiotherapy
  The incidence of radiation pneumonia
Percentage of subjects with radiation pneumonia of ≥ Grade 3 | up to 24 weeks after completion of radiotherapy
  Percentage of subjects with radiation pneumonia of ≥ Grade 3 evaluated by CTCAE v5.0
Severity at the first diagnosis of radiation pneumonia | up to 24 weeks after completion of radiotherapy
  Severity at the first diagnosis of radiation pneumonia evaluated by CTCAE v5.0
Maximum severity of radiation pneumonia | up to 24 weeks after completion of radiotherapy
  Maximum severity of radiation pneumonia evaluated by CTCAE v5.0
Changes in lung function | at 4 weeks and 12 weeks after completion of radiotherapy
  Changes in lung function (FEV1, DL CO) at each time point after administration compared to before administration of investigational products
The incidence of pulmonary fibrosis | at 24 weeks after completion of radiotherapy
  The incidence of pulmonary fibrosis
Lung fibrosis area | at 24 weeks after completion of radiotherapy
  Lung fibrosis area
Lung volume reduction | at 24 weeks after completion of radiotherapy
  Lung volume reduction
Pulmonary toxicity grade | at the time of initial diagnosis of radiation pneumonia after completion of radiotherapy
  Pulmonary toxicity grade evaluated by Radiation Therapy Oncology Group (RTOG) Acute radiation morbidity
The maximum grade of lung toxicity | up to 24 weeks after completion of radiotherapy
  The maximum grade of lung toxicity evaluated by RTOG Acute radiation morbidity

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea